CLINICAL TRIAL: NCT05725772
Title: Comparison of Different Health Care Delivery Methods in a Rural Underserved Population of People With Parkinson's Disease
Brief Title: Comparison of Health Care Delivery Methods in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 274510
Record Dates: First submitted 2023-02-03; First posted 2023-02-13 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: medically underserved areas; telemedicine; remote monitoring
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease: People with Parkinson's disease living in medically underserved areas
  Interventions: Other: Location of Visit

INTERVENTIONS:
Other: Location of Visit — Participants will perform visits 1) at-home via telemedicine, 2) in-person and 3) at a local regional clinic via telemedicine

SUMMARY:
The goal of this observational study is to compare the ability to perform telemedicine visits at home, at a regional clinic close to home, and in-person in People with Parkinson's disease. The main question it aims to answer is whether telemedicine assessments provide high quality care to people with Parkinson's disease. Participants will perform a regular clinic visit followed by research evaluations of their disease. Researchers will compare the results of these assessments at the different visit types to see if there are differences in the results.

DETAILED DESCRIPTION:
The purpose of the current project is to determine whether care for people with Parkinson's disease can be performed as well using telemedicine as it can be when people visit their neurologist in-person. We hope that the findings from this project will help 1) improve the quality and access of healthcare to those parts of Arkansas where access may be limited, 2) decrease the costs of healthcare in movement disorders, and 3) allow more people with Parkinson's disease to feel like they are participating in finding a cure by taking part in research. It will also allow us to improve on ways to collect information from people with Parkinson's, even in their own homes, to help us design future research studies. This will be important to help develop treatments that are for each person, not just the disease as a whole.

Specific Aims of the Study:

AIM 1: To determine whether telehealth assessments provide high quality care to people with Parkinson's disease. We will do this by performing and comparing the results of assessments that are regularly used in clinics and in research repeated in 3 different settings, at-home via telehealth, at a regional center via telehealth, and in-person at UAMS.

AIM 2: To improve tools for studying large collections of information that are collected using multiple different methods. We will do this by using a health information database that we have developed for this purpose. We will use voice and handwriting analysis compared in the three different settings to develop ways to track disease progression in Parkinson's disease.

How we plan to accomplish those Aims:

All people with Parkinson's who agree to participate will have their regular clinical visits with Dr. Tuhin Virmani or Dr. Rohit Dhall at home and at a UAMS regional clinic center near their homes. Following the clinic portion of the visit they will provide a sample of their speech and handwriting, undergo a timed walk, have their thinking ability tested, and fill out some questionnaires and surveys about their mood, anxiety, quality of life, and sleep quality. They will also be asked to complete surveys to allow us to determine who they feel the quality of each visit type was and at the end compare one to the other. These different sources of information from each person will then be combined together and stored in our database, and used by the research team to develop new tools to combine and compare such different types of information to better treat people with Parkinson's Disease in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 45- to 90-years old
* Diagnosis of idiopathic PD as defined by the UK Brain Bank criteria.

Exclusion Criteria:

* Cognitive impairments sufficient to preclude capacity to provide informed consent, as determined by Dr. Virmani or Dr. Dhall on the basis of each potential participant's stated understanding of the study following review of the consent form;
* Diagnosis of neurological disorder other than PD
* Diagnosis of a psychiatric disorder (other than depression or anxiety from PD)
* Use of anti-dopaminergic medications in 1-year period prior to enrollment
* Inability to complete questionnaires or effectively communicate in English
* Inability to perform research assessments via smartphone, tablet or computer.

Ages: 45 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's disease living in designated medically underserved areas.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of remote data collection | 12 weeks
  Feasibility of remotely collecting high-quality research data on a smartphone, tablet, or home computer.

CONTACTS AND LOCATIONS:
Overall Officials: Tuhin Virmani, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No